CLINICAL TRIAL: NCT00737477
Title: A Single Arm, Open-Label, Multicentre Study to Assess the Maintenance of Haemoglobin Levels With Once Monthly Subcutaneous Administration of C.E.R.A (Continuous Erythropoietin Receptor Activator) in Patients With Chronic Kidney Disease on Peritoneal Dialysis
Brief Title: A Study of Monthly Subcutaneous (SC) Mircera for Maintenance Treatment of Participants With Chronic Kidney Disease on Peritoneal Dialysis
Acronym: MISTRAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21421; 2008-001747-18 (EudraCT Number)
Record Dates: First submitted 2008-08-18; First posted 2008-08-19 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-05

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

ARMS (1):
- Mircera in Renal Anemia (Experimental): Participants will receive SC methoxy polyethylene glycol-epoetin beta (Mircera) every 4 weeks for a total of 48 weeks in this single-arm study. The first dose of 120 or 200 micrograms (mcg) will be determined by the dose of ESA received prior to administration of study treatment, while subsequent doses will be adjusted to maintain hemoglobin within the target range.
  Interventions: Drug: Methoxy polyethylene glycol-epoetin beta

INTERVENTIONS:
Drug: Methoxy polyethylene glycol-epoetin beta — Mircera will be administered SC every 4 weeks for a total of 48 weeks. The first dose of 120 or 200 mcg will be determined by the dose of ESA received prior to administration of study treatment, while subsequent doses will be adjusted to maintain hemoglobin within the target range.
  Other Names: Mircera; CERA

SUMMARY:
This single-arm study will assess the efficacy and safety of monthly administration of SC Mircera for the maintenance of hemoglobin levels in participants with chronic kidney disease on peritoneal dialysis. Participants currently receiving maintenance treatment with SC erythropoietin stimulating agents (ESAs) will receive monthly SC injections of Mircera, with the starting dose derived from the last weekly ESA they had been receiving.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than or equal to (≥) 18 years of age
* Chronic kidney disease-related anemia on peritoneal dialysis for ≥3 months
* Continuous SC maintenance stable ESA therapy for 4 weeks prior to study start

Exclusion Criteria:

* Transfusion of red blood cells during previous 8 weeks
* Poorly controlled hypertension requiring interruption of ESA treatment in previous 6 months
* Significant acute or chronic bleeding during previous 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2008-09-30 (Actual); Primary Completion 2011-07-31 (Actual); Study Completion 2011-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (52):
- France (52):
  - Ch Notre Dame Misericorde; Hemodialyse, Ajaccio
  - Centre Hospitalier; Hemodialyse, Annonay
  - Ch D Arras; Nephrologie, Arras
  - Ch D Auxerre; Nephrologie Hemodialyse, Auxerre
  - CHU Saint Jacques; Centre De Dialyse, Besançon
  - Ch Germon Et Gauthier; Hemodialyse, Beuvry
  - Polyclin Bordeaux Nord Aquitaine; Nephrologie - Hemodialyse, Bordeaux
  - Centre D Hemodialyse Saint Roch, Cabestany
  - Hopital Clemenceau; Nephrologie Hemodialyse, Caen
  - Hôpital Des Brousailles; Service de Néphrologie, Cannes
  - CH William Morey; Nephrologie, Chalon-sur-Saône
  - Ch De Chambery; Nephrologie, Chambéry
  - Hopital Manchester; Nephrologie Hemodialyse, Charleville-Mézières
  - Ch Hotel Dieu; Nephrologie, Chartres
  - Ch Du Cotentin Site De Cherbourg; Nephrologie, Cherbourg Octeville
  - Hopital Louis Pasteur; Nephrologie - Hemodialyse, Colmar
  - Ch Laennec; Nephrologie Hemodialyse, Creil
  - Hopital Du Bocage; Nephrologie, Dijon
  - Ch De Dunkerque; Nephrologie, Dunkirk
  - Chi Eure Seine D Evreux; Nephrologie, Évreux
  - Agduc Muller, La Tronche
  - Anider; Pharmacie, Le Petit-Quevilly
  - Hopital Calmette; Medecine General & Nephrologie Serv., Lille
  - Ch Robert Bisson; Nephrologie, Lisieux
  - Aural, Lyon
  - Hopital Marc Jacquet; Nephrologie Hemodialyse, Melun
  - Hopital Saint Andre; Nephrologie, Metz
  - Echo Nantes Confluent; Uad Montfort, Nantes
  - Ch Georges Renon; Nephrologie Hemodialyse, Niort
  - Hopital de La Source; Service de Nephrologie & Hemodialyse, Orléans
  - Unite Autodialyse Paris 14; Dialyse A Domicile, Paris
  - Ch Pitie Salpetriere; Nephrologie Hemodialyse, Paris
  - Hopital Bichat Claude Bernard; Nephrologie, Paris
  - Hopital Tenon; Nephrologie Dialyse, Paris
  - Chu La Miletrie;Nephrologie Transplantation, Poitiers
  - Ch Rene Dubos; Dialyse Peritoneale, Pontoise
  - Chi De Cornouaille; Nephrologie, Quimper
  - Hopital De La Maison Blanche; Nephrologie Hemodialyse, Reims
  - Ch De Bourran; Nephrologie Hemodialyse, Rodez
  - Aurar; Aurar St Denis, Saint-Denis
  - Memorial France Etats Unis; Nephrologie, Saint-Lô
  - Hopital National; Nephrologie Hemodialyse, Saint-Maurice
  - Aurar, Saint-Pierre
  - HOPITAL NORD; NEPH Transplantation Reanimation, Saint-Priest-en-Jarez
  - CH de Saintonge; Unite 1 Med Interne Nephrologie, Saintes
  - Ch De Soissons; Medecine 5, Soissons
  - Hopital Civil; Nephrologie Clinique Medicale B, Strasbourg
  - Arauco; Arauco Tours Bretonneau, Tours
  - Ch De Valence; Departement Medecine, Valence
  - ALTIR, Vandœuvre-lès-Nancy
  - CH Bretagne Atlantique de Vannes; Hemodialyse, Vannes
  - Ch De Vittel; Nephrologie Hemodialyse, Vittel

RESULTS

PARTICIPANT FLOW:
Groups:
- Mircera in Chronic Kidney Disease (CKD)-Related Anemia: Participants with CKD-related anemia undergoing peritoneal dialysis and who were previously treated with erythropoiesis-stimulating agent (ESA) therapy received subcutaneous (SC) methoxy polyethylene glycol-epoetin beta (Mircera), also known as continuous erythropoietin receptor activator (CERA), every 4 weeks in this single-arm study. The first dose of 120 or 200 micrograms (mcg) during Week 0 was based upon the dose of ESA received during the initial 4-week screening period, while subsequent doses were adjusted from Weeks 4 to 12 during the dose adaptation period (DAP) to maintain target hemoglobin (Hb) concentrations within 10 to 12 grams per deciliter (g/dL). Treatment continued during a designated efficacy evaluation period (EEP) from Weeks 16 to 24 and an additional follow-up period from Weeks 28 to 48.
Period: Overall Study
Arm/Group | Mircera in Chronic Kidney Disease (CKD)-Related Anemia
Started | 96
Completed | 62
Not Completed | 34
Not completed — Adverse Event | 9
Not completed — Death | 9
Not completed — Treatment Refusal | 1
Not completed — Withdrawal by Subject | 1
Not completed — Renal Transplantation | 10
Not completed — Other | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who received at least one dose of Mircera and provided at least one Hb evaluation between Weeks 0 to 24, and for whom any follow-up information was available.
Groups:
- Mircera in CKD-Related Anemia: Participants with CKD-related anemia undergoing peritoneal dialysis and who were previously treated with ESA therapy received SC Mircera/CERA every 4 weeks in this single-arm study. The first dose of 120 or 200 mcg during Week 0 was based upon the dose of ESA received during the initial 4-week screening period, while subsequent doses were adjusted from Weeks 4 to 12 during the DAP to maintain target Hb concentrations within 10 to 12 g/dL. Treatment continued during a designated EEP from Weeks 16 to 24 and an additional follow-up period from Weeks 28 to 48.
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Maintained Average Hb Value Within Target Range During the EEP
Description: Participants provided pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. The average Hb during the EEP (Weeks 16 to 24) was calculated per participant and assessed against the target range. The percentage of participants who had average Hb during the EEP in the target range (10 to 12 g/dL) was determined as the primary endpoint. The 95 percent (%) confidence interval (CI) was calculated using the Pearson-Clopper method for exact confidence bounds.
Time Frame: Weeks 16 to 24
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided sufficient data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 80
percentage of participants | 50.0 [39.0 to 61.0]

2. Secondary Outcome: Percentage of Participants With Hb Values Within Target Range During the EEP
Description: During the EEP (Weeks 16 to 24), participants provided a total of three pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. The percentage of participants who had at least one, two, or all three Hb values during the EEP in the target range (10 to 12 g/dL) was determined.
Time Frame: Weeks 16 to 24
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided sufficient data for at least one Hb value. The number of participants who provided sufficient data for each analysis (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 80
percentage of participants
  At Least One Hb Value (n=80) | 78.8
  At Least Two Hb Values (n=77) | 49.4
  All Three Hb Values (n=74) | 23.0

3. Secondary Outcome: Change in Hb Value From Baseline to the EEP
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment screening period (Weeks -4 to 0). Participants provided pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. The average Hb during the EEP (Weeks 16 to 24) was calculated per participant and assessed against the reference value. The mean change in Hb value between reference (i.e., "Baseline") Hb and the EEP average Hb was calculated and expressed in g/dL.
Time Frame: Baseline and Weeks 16 to 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 80
g/dL | 0.4 (0.9)

4. Secondary Outcome: Time Spent in the Target Range for Hb During the EEP and the Overall Treatment Period
Description: Participants provided pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Time spent in the target range (10 to 12 g/dL) was defined as time from first on-target Hb measurement to time of last known on-target Hb measurement, as collected during the EEP (Weeks 16 to 24) and the overall treatment period (Weeks 0 to 48). Time spent in the target range was averaged among all participants and expressed in weeks.
Time Frame: Weeks 16 to 24 and Weeks 0 to 48
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided sufficient data. The number of participants who provided sufficient data within each timeframe (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 94
weeks
  EEP (Weeks 16 to 24; n=80) | 5.9 (4.2)
  Overall Study (Weeks 0 to 48; n=94) | 22.0 (13.8)

5. Secondary Outcome: Percentage of Participants With Hb Value Within Plus/Minus (±) 1 g/dL of Reference Hb and Within the Target Range by Study Visit
Description: Reference Hb was determined individually per participant as the average of all Hb values during a pre-treatment screening period (Weeks -4 to 0). Participants provided pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. The percentage of participants who had average Hb during the EEP (Weeks 16 to 24) and follow-up (Weeks 28 to 48) in the target range (10 to 12 g/dL) and within ±1 g/dL of their individual reference Hb was determined by study visit.
Time Frame: Baseline and Weeks 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided sufficient data. The number of participants who provided sufficient data at each timepoint (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
percentage of participants
  Week 16 (n=80) | 37.5
  Week 20 (n=76) | 35.5
  Week 24 (n=75) | 44.0
  Week 28 (n=73) | 39.7
  Week 32 (n=72) | 44.4
  Week 36 (n=68) | 51.5
  Week 40 (n=65) | 44.6
  Week 44 (n=63) | 44.4
  Week 48 (n=62) | 38.7

6. Secondary Outcome: Percentage of Participants With Cycles or Excursions
Description: Participants provided pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA. Cycles were defined as a change in Hb greater than (>) 1.5 g/dL lasting longer than 8 weeks. Excursions were defined as half of one full cycle, or an increase ("up" excursions) or decrease ("down" excursions) >1.5 g/dL lasting longer than 4 weeks according to Hb measurements collected during the study. The percentage of participants with at least one cycle or excursion during Weeks 4 to 44 was calculated.
Time Frame: Weeks 4 to 44
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
percentage of participants
  At Least One Cycle | 5.3
  At Least One Excursion | 60.0
  At Least One Up Excursion | 46.3
  At Least One Down Excursion | 18.9

7. Secondary Outcome: Percentage of Participants With Up Excursions
Description: Participants provided pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA during the DAP, EEP, and follow-up. Excursions were defined as half of one full cycle, or an increase ("up" excursions) or decrease ("down" excursions) in Hb >1.5 g/dL lasting longer than 4 weeks. The percentage of participants with at least one up excursion was calculated for Weeks 4 to 16, Weeks 16 to 24, and Weeks 24 to 44.
Time Frame: Weeks 4 to 16, Weeks 16 to 24, Weeks 24 to 44
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants with at least one up excursion.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 44
percentage of participants
  Weeks 4 to 16 | 31.8
  Weeks 16 to 24 | 45.5
  Weeks 24 to 44 | 22.7

8. Secondary Outcome: Percentage of Participants With Down Excursions
Description: Participants provided pre-dose blood samples for Hb monitoring while on treatment with Mircera/CERA during the DAP, EEP, and follow-up. Excursions were defined as half of one full cycle, or an increase ("up" excursions) or decrease ("down" excursions) in Hb >1.5 g/dL lasting longer than 4 weeks. The percentage of participants with at least one down excursion was calculated for Weeks 4 to 16, Weeks 16 to 24, and Weeks 24 to 44.
Time Frame: Weeks 4 to 16, Weeks 16 to 24, Weeks 24 to 44
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants with at least one down excursion.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 18
percentage of participants
  Weeks 4 to 16 | 16.7
  Weeks 16 to 24 | 11.1
  Weeks 24 to 44 | 72.2

9. Secondary Outcome: Percentage of Participants Who Required Any Dose Adjustment of Mircera/CERA
Description: Study drug administration occurred monthly during treatment (Weeks 0 to 48), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during the initial 4-week screening period. Subsequent doses could be adjusted on the basis of Hb levels or other modification criteria. The percentage of participants who required any dose adjustment (including decreased dose, increased dose, and dose not performed) was calculated for Weeks 4 to 20, Weeks 24 to 48, and Weeks 4 to 48.
Time Frame: Weeks 4 to 20, Weeks 24 to 48, Weeks 4 to 48
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided sufficient data. The number of participants who provided sufficient data for each analysis within each timeframe (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
percentage of participants
  Any Dose Adjustment, Weeks 4 to 20 (n=95) | 84.2
  Decreased Dose, Weeks 4 to 20 (n=75) | 69.3
  Increased Dose, Weeks 4 to 20 (n=75) | 43.3
  Dose Not Performed, Weeks 4 to 20 (n=95) | 34.7
  Any Dose Adjustment, Weeks 24 to 48 (n=76) | 100
  Decreased Dose, Weeks 24 to 48 (n=50) | 74.0
  Increased Dose, Weeks 24 to 48 (n=50) | 46.0
  Dose Not Performed, Weeks 24 to 48 (n=76) | 30.3
  Any Dose Adjustment, Weeks 4 to 48 (n=95) | 96.8
  Decreased Dose, Weeks 4 to 48 (n=94) | 84.0
  Increased Dose, Weeks 4 to 48 (n=94) | 71.3
  Dose Not Performed, Weeks 4 to 48 (n=95) | 47.4

10. Secondary Outcome: Number of Dose Adjustments of Mircera/CERA
Description: Study drug administration occurred monthly during treatment (Weeks 0 to 48), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during the initial 4-week screening period. Subsequent doses could be adjusted on the basis of Hb levels or other modification criteria. The number of dose adjustments performed for each participant was averaged among all participants for Weeks 4 to 20, Weeks 24 to 48, and Weeks 4 to 48.
Time Frame: Weeks 4 to 20, Weeks 24 to 48, Weeks 4 to 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: dose adjustments
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
dose adjustments
  Weeks 4 to 20 (n=95) | 2.0 (1.3)
  Weeks 24 to 48 (n=76) | 5.6 (1.3)
  Weeks 4 to 48 (n=95) | 3.3 (2.0)

11. Secondary Outcome: Absolute Change in Dose of Mircera/CERA by Study Week
Description: Study drug administration occurred monthly during treatment (Weeks 0 to 48), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during the initial 4-week screening period. Subsequent doses could be adjusted on the basis of Hb levels or other modification criteria. The absolute difference in dose from the previous week was calculated at each visit and averaged among all participants.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: ITT Population. The "Number of Participants Analyzed" reflects the total number of participants who provided sufficient data. The number of participants who provided sufficient data for each analysis at each timepoint (n) is shown in the table.
Measure: Mean (Standard Deviation); unit: mcg
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
mcg
  Week 4, Dose Decrease (n=25) | 25.8 (11.9)
  Week 4, Dose Increase (n=9) | 37.8 (17.2)
  Week 8, Dose Decrease (n=32) | 28.4 (12.3)
  Week 8, Dose Increase (n=14) | 42.9 (24.6)
  Week 12, Dose Decrease (n=21) | 24.5 (3.5)
  Week 12, Dose Increase (n=8) | 52.5 (21.7)
  Week 16, Dose Decrease (n=20) | 24.0 (2.6)
  Week 16, Dose Increase (n=8) | 47.5 (29.0)
  Week 20, Dose Decrease (n=11) | 29.1 (15.3)
  Week 20, Dose Increase (n=10) | 34.5 (11.2)
  Week 24, Dose Decrease (n=18) | 29.0 (12.2)
  Week 24, Dose Increase (n=10) | 50.5 (26.0)
  Week 28, Dose Decrease (n=13) | 38.5 (22.0)
  Week 28, Dose Increase (n=7) | 35.0 (20.2)
  Week 32, Dose Decrease (n=10) | 27.0 (8.8)
  Week 32, Dose Increase (n=8) | 37.5 (19.1)
  Week 36, Dose Decrease (n=10) | 28.5 (11.6)
  Week 36, Dose Increase (n=2) | 75.0 (35.4)
  Week 40, Dose Decrease (n=11) | 37.3 (26.8)
  Week 40, Dose Increase (n=4) | 22.5 (2.9)
  Week 44, Dose Decrease (n=2) | 18.5 (2.1)
  Week 44, Dose Increase (n=5) | 32.0 (10.9)
  Week 48, Dose Decrease (n=0) | NA (NA) — No dose decreases were performed at the designated visit.
  Week 48, Dose Increase (n=2) | 40.0 (14.1)

12. Secondary Outcome: Percent Change in Dose of Mircera/CERA by Study Week
Description: Study drug administration occurred monthly during treatment (Weeks 0 to 48), which began with a pre-specified dose of Mircera/CERA according to the dose of ESA administered during the initial 4-week screening period. Subsequent doses could be adjusted on the basis of Hb levels or other modification criteria. The percent difference in dose from the previous week was calculated at each visit as [(current dose minus previous week dose) divided by previous week dose] multiplied by 100, and averaged among all participants.
Time Frame: Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: percent change in dose
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
percent change in dose
  Week 4, Dose Decrease (n=25) | 23.7 (9.0)
  Week 4, Dose Increase (n=9) | 22.2 (6.7)
  Week 8, Dose Decrease (n=32) | 33.3 (22.2)
  Week 8, Dose Increase (n=14) | 21.4 (4.9)
  Week 12, Dose Decrease (n=21) | 30.3 (10.0)
  Week 12, Dose Increase (n=8) | 22.0 (2.3)
  Week 16, Dose Decrease (n=20) | 41.1 (14.0)
  Week 16, Dose Increase (n=8) | 25.6 (7.7)
  Week 20, Dose Decrease (n=11) | 57.6 (60.7)
  Week 20, Dose Increase (n=10) | 21.5 (4.6)
  Week 24, Dose Decrease (n=18) | 45.0 (24.8)
  Week 24, Dose Increase (n=10) | 29.6 (14.5)
  Week 28, Dose Decrease (n=13) | 38.5 (12.0)
  Week 28, Dose Increase (n=7) | 29.7 (7.1)
  Week 32, Dose Decrease (n=10) | 36.5 (16.4)
  Week 32, Dose Increase (n=8) | 24.6 (6.2)
  Week 36, Dose Decrease (n=10) | 43.7 (15.5)
  Week 36, Dose Increase (n=2) | 22.5 (3.5)
  Week 40, Dose Decrease (n=11) | 51.6 (29.3)
  Week 40, Dose Increase (n=4) | 26.7 (9.7)
  Week 44, Dose Decrease (n=2) | 35.8 (22.3)
  Week 44, Dose Increase (n=5) | 24.0 (8.9)
  Week 48, Dose Decrease (n=0) | NA (NA) — No dose decreases were performed at the designated visit.
  Week 48, Dose Increase (n=2) | 22.5 (3.5)

13. Secondary Outcome: Percentage of Participants Requiring Blood Transfusions
Description: The percentage of participants who received at least one red blood cell transfusion during the overall treatment period (Weeks 0 to 48) was calculated.
Time Frame: Weeks 0 to 48
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Mircera in CKD-Related Anemia
Number analyzed (Participants) | 95
percentage of participants | 3.2

ADVERSE EVENTS:
Time Frame: Continuously from Weeks -4 to 48 and/or 30 days after last dose (up to approximately 1 year overall)
Description: Safety Population: All participants who received at least one dose of Mircera and for whom any follow-up information was available.
Arm/Group | Mircera in CKD-Related Anemia
Serious Adverse Events (participants affected / at risk) | 48/96
Other Adverse Events (participants affected / at risk) | 25/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in CKD-Related Anemia (N=96)
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal polyp (Gastrointestinal disorders) | 1
Oesophagitis haemorrhagic (Gastrointestinal disorders) | 1
Oesophagitis ulcerative (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Peritonitis (Gastrointestinal disorders) | 7
Pneumoperitoneum (Gastrointestinal disorders) | 1
Subileus (Gastrointestinal disorders) | 1
Umbilical hernia (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Acute coronary syndrome (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrioventricular block (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure acute (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Laryngitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Peritoneal candidiasis (Infections and infestations) | 1
Peritoneal infection (Infections and infestations) | 3
Sepsis (Infections and infestations) | 2
Asthenia (General disorders) | 1
General physical health deterioration (General disorders) | 2
Hyperthermia (General disorders) | 1
Oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Product contamination microbial (General disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Coma (Nervous system disorders) | 1
Convulsion (Nervous system disorders) | 1
Mental impairment (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Arterial disorder (Vascular disorders) | 1
Extremity necrosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 2
Thrombosis (Vascular disorders) | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholecystitis acute (Hepatobiliary disorders) | 2
Clavicle fracture (Musculoskeletal and connective tissue disorders) | 1
Femoral neck fracture (Musculoskeletal and connective tissue disorders) | 1
Spinal compression fracture (Musculoskeletal and connective tissue disorders) | 1
Macular oedema (Eye disorders) | 1
Post procedural complication (Injury, poisoning and procedural complications) | 1
Blood glucose fluctuation (Investigations) | 1
Confusional state (Psychiatric disorders) | 1
Removal of ambulatory peritoneal catheter (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Mircera in CKD-Related Anemia (N=96)
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 5
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 11
Hypertension (Vascular disorders) | 8
Oedema peripheral (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.